CLINICAL TRIAL: NCT04246983
Title: Introducing Point-of-care Ultrasound at the Bedside for Diagnosing Opportunistic Diseases in Patients With HIV
Brief Title: Point-of Care Ultrasound for Patients With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Mischa Huson, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL72666.078.20
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS; Opportunistic Infections, HIV Related
Keywords: HIV; Opportunistic disease; Ultrasound
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; AIDS-Related Opportunistic Infections | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HIV undergoing point of care ultrasound (Experimental)
  Interventions: Diagnostic Test: Opportunistic infection Ultrasound (OpUS) screening

INTERVENTIONS:
Diagnostic Test: Opportunistic infection Ultrasound (OpUS) screening — this point-of-care ultrasound protocol will include lung ultrasound, assessment of pericardial and pleural effusions, ascites, abdominal lymphadenopathy and splenic micro abscesses, as well as a focused ultrasound of liver and kidneys.

SUMMARY:
Rationale: Point-of-care ultrasound (POCUS) is increasingly used by various specialists in the Netherlands, but its role in managing patients with HIV is unclear. In settings endemic for tuberculosis, Fast Assessment with Sonography for HIV/Tuberculosis (FASH) has proven its value to detect extrapulmonary tuberculosis in patients with HIV. However, there is no data to support POCUS for patients with HIV in resource affluent settings.

Objective: The investigators aim to determine the feasibility and diagnostic value of POCUS in detecting opportunistic disease in HIV patients with advanced disease stages in the Netherlands.

Study design: The investigators will perform a prospective observational pilot study.

Study population: The investigators will include new adult patients with HIV presenting with a cluster of differentiation 4 (CD4) T-cell count below 350 cells/mm3, and all adult HIV patients requiring admission to hospital. Intervention (if applicable): The investigators will perform a focused ultrasound examination including FASH, and ultrasound of the lung, liver and kidneys. In case of positive findings additional examinations will be undertaken to determine the underlying pathology and/or treatment started as indicated. In case of negative findings, patients will be followed for 12 months to observe for (possibly missed) opportunistic infections.

Main study parameters/endpoints: Our primary outcomes include acceptability of POCUS by patients, interobserver variation in interpretation of POCUS images, and number of diagnosed AIDS and non-AIDS related problems. Secondary outcomes include sensitivity and specificity, negative predictive value and positive predictive value of our POCUS protocol. In addition, incidence rates of opportunistic infections will be compared to a historical matched control group.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The ultrasound examination is painless and without risk to the participants. It will take approximately 30 minutes and will be combined with routine visits to the hospital. Benefits include potential earlier detection of opportunistic disease, while adverse effects may arise from false positive findings requiring further examinations which may cause stress or anxiety. The rate of false positive findings in POCUS has not been formally investigated, but appears low. The effect of POCUS in advanced HIV/AIDS can only be studied in HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* new patients with HIV presenting with a CD4 T-cell count below 350 cells/mm3
* patients with HIV who are admitted to hospital

Exclusion Criteria:

- absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of point-of-care ultrasound by patients | 1 day
interobserver variation in interpretation of ultrasound images | 1 day
Number of diagnosed AIDS and non-AIDS related problems | 1 year

SECONDARY OUTCOMES:
Sensitivity and specificity, negative predictive value and positive predictive value of our ultrasound protocol to diagnose opportunistic disease. | 1 year
Number of diagnosed AIDS and non-AIDS related problems compared to a historic control group | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mischa Huson, MD, PhD, Principal Investigator — Erasmus Medical Centre
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heller T, Wallrauch C, Goblirsch S, Brunetti E. Focused assessment with sonography for HIV-associated tuberculosis (FASH): a short protocol and a pictorial review. Crit Ultrasound J. 2012 Nov 21;4(1):21. doi: 10.1186/2036-7902-4-21. PMID 23171481
- [Background] Heller T, Mtemang'ombe EA, Huson MA, Heuvelings CC, Belard S, Janssen S, Phiri S, Grobusch MP. Ultrasound for patients in a high HIV/tuberculosis prevalence setting: a needs assessment and review of focused applications for Sub-Saharan Africa. Int J Infect Dis. 2017 Mar;56:229-236. doi: 10.1016/j.ijid.2016.11.001. Epub 2016 Nov 9. PMID 27836795
- [Background] Giordani MT, Tamarozzi F, Kaminstein D, Brunetti E, Heller T. Point-of-care lung ultrasound for diagnosis of Pneumocystis jirovecii pneumonia: notes from the field. Crit Ultrasound J. 2018 Apr 17;10(1):8. doi: 10.1186/s13089-018-0089-0. PMID 29666966
- [Background] Hunter L, Belard S, Janssen S, van Hoving DJ, Heller T. Miliary tuberculosis: sonographic pattern in chest ultrasound. Infection. 2016 Apr;44(2):243-6. doi: 10.1007/s15010-015-0865-8. Epub 2015 Dec 11. PMID 26661658
- [Background] Agostinis P, Copetti R, Lapini L, Badona Monteiro G, N'Deque A, Baritussio A. Chest ultrasound findings in pulmonary tuberculosis. Trop Doct. 2017 Oct;47(4):320-328. doi: 10.1177/0049475517709633. Epub 2017 May 25. PMID 28541140
- [Background] Giordani MT, Brunetti E, Binazzi R, Benedetti P, Stecca C, Goblirsch S, Heller T. Extrapulmonary mycobacterial infections in a cohort of HIV-positive patients: ultrasound experience from Vicenza, Italy. Infection. 2013 Apr;41(2):409-14. doi: 10.1007/s15010-012-0336-4. Epub 2012 Sep 24. PMID 23001543
- [Background] Schouten M, van Velde AJ, Snijdewind IJ, Verbon A, Rijnders BJ, van der Ende ME. [Late diagnosis of HIV positive patients in Rotterdam, the Netherlands: risk factors and missed opportunities]. Ned Tijdschr Geneeskd. 2013;157(15):A5731. Dutch. PMID 23575291
- [Background] French MA, Price P, Stone SF. Immune restoration disease after antiretroviral therapy. AIDS. 2004 Aug 20;18(12):1615-27. doi: 10.1097/01.aids.0000131375.21070.06. PMID 15280772
- [Derived] Huson M, Rokx C. Exploring the role of point-of-care ultrasound for people with HIV in a resource affluent setting: A prospective observational study. Int J STD AIDS. 2023 Nov;34(13):984-989. doi: 10.1177/09564624231188744. Epub 2023 Jul 27. PMID 37500120